CLINICAL TRIAL: NCT01056861
Title: Effects of Botulinum on the Afferent Input Modulation of Neuronal Circuits Involved in Cervical Dystonia
Brief Title: Effects of Botulinum Toxin in Cervical Dystonia
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Naganad Sripathi, Senior Staff Neurologist, Henry Ford Health System
Other Study IDs: 5307; 08-0124 (Other Grant/Funding Number: Allergan1)
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Torticollis; Cervical Dystonia
Keywords: cervical dystonia; torticollis; Botulinum toxin; magnetoencephalography; MEG; cortical organizational changes detected by MEG after botulinum toxin in patients with torticollis, correlating with improvement in the symptoms
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cervical dystonia (torticollis): Subjects meeting the criteria fot torticollis who are receiving botulinum toxin injections.
  Interventions: Drug: Botulinum Toxin A
- Control: age matched controls with out cervical dystonia (torticollis)
  Interventions: Drug: Botulinum Toxin A

INTERVENTIONS:
Drug: Botulinum Toxin A — Not exceeding a total dose of 400 units, once every three months.
  Other Names: Botox, Botulinum toxin A

SUMMARY:
Botulinum toxin injection in the contracting muscles has proven to be a safe and effective method of relieving pain and lessening dystonic posturing. The current hypothesis is that botulinum toxin works on altering sensory input in the central nervous system in addition to its effects on the neuromuscular junction.

Magnetoencephalography (MEG)of brain has been used in dystonia such as writer's cramp and musician's hand dystonia. However, no study has investigated the correlation of central signal changes via magnetoencephalography before and after treatment with botulinum in torticollis patients. Prior studies using somatosensory potentials indicated the possibility of differential activation of precentral cortex in patients with cervical dystonia. Cervical dystonia may result from a disorder of both cortical excitability and intracortical inhibition. The investigators hypothesis is that botulinum injection modulates central inhibition which improves clinical outcome for torticollis.

DETAILED DESCRIPTION:
This study of MEG neuro-imagery will increase the understanding of the central pathway involvement in the efficacy of botulinum toxin treatment for torticollis. Cervical dystonia (spasmodic torticollis) patients will be selected from the Neurology clinic. Subjects will range in age from 18 years old through 90 years old. Subjects are expected to be ambulatory and independent. Patients are generally expected to be in good health. Exclusion criteria include significant intracranial metal (typically fixed dental bridges or braces) generating significant magnetic artifact, medical instability, pregnancy, and certain other factors such as severe head tremors that would produce magnetic artifact. Clinical states of torticollis patients will be assessed by using Tsui scale. Every torticollis patient will have magnetoencephalography on the day of botulinum treatment beforehand and approximately 2-8 weeks after botulinum treatment. We will compare the results of magnetoencephalography between control subject and torticollis patient before botulinum treatment aiming to find any difference between the two populations. We also compare the results of magnetoencephalography in individual torticollis patient before and after botulinum treatment, aiming to detect the changes between these two conditions in the same individual and possibly between the average of data from each condition before and after botulinum treatment.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects 18 years to 90 years
* females who are child bearing potential, with negative pregnancy testing, who are willing to use reliable form of contraception during the study
* subjects meeting the criteria for torticollis

Exclusion Criteria:

* intracranial metal objects generating significant magnetic artifact
* females who are pregnant, planning pregnancy, unable to use contraception
* mental instability
* any medical condition that may put the subject at increased risk with exposure to botulinum toxin, allergy or sensitivity
* significant head tremor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects meeting the criteria for cervical dystonia (torticollis) who are receiving botulinum toxin injections in the Neurology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evidence of Cortical organizational changes with botulinum toxin treatment in patients with torticollis utilizing magnetoencephalography | two to eight weeks following treatment

SECONDARY OUTCOMES:
Tsui Torticollis Rating scale | Two-eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Naganand Sripathi, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States